CLINICAL TRIAL: NCT05023850
Title: Comparing Thoracolumbar Interfascial Plane Block With Erector Spinae Plane Block for Thoracolumbar Decompressive Surgery: a Randomized Clinical Trial
Brief Title: Comparing Thoracolumbar Interfascial Plane Block With Erector Spinae Plane Block
Acronym: TLIPvsESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-2021/13
Record Dates: First submitted 2021-08-19; First posted 2021-08-27 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-09

CONDITIONS: Spinal Surgery; Quality of Recovery; Postoperative Analgesia; Postoperative Complications
Keywords: Thoracolumbar Interfascial Plane Block; Erector Spinae Plane Block; Thoracolumbar Decompressive Surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomized control trial one group receives Thoracolumbar Interfascial Plane Block the other receives Erector Spinae Plane Block
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blocks will be administered after induction of General Anesthesia so participants will be blinded to which intervention they have had.
  Study investigators will not be aware of what group the participant belongs to when assessing the patient's post-operative period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TLIP (Active Comparator): Patients will receive a Thoracolumbar Plane Block (TLIPB) under ultrasound guidance while under general anesthesia.
  Intervention: Patients will receive a TLIPB with 20mls 0.25% Bupivicaine bilaterally.
  Interventions: Procedure: TLIPB
- Group ESP (Experimental): Patients will receive an Erector Spinae Plane Block (ESPB) under ultrasound guidance while under general anesthesia.
  Intervention: Procedure: Patients will receive an ESPB with 20 ml 0.25% Bupivacaine bilaterally.
  Interventions: Procedure: ESPB

INTERVENTIONS:
Procedure: TLIPB — Patients will receive TLIPB with an injection of 40 ml of bupivacaine 0.25% (2 injections of 20 ml on each side) between multifidus and longissimus muscles.
  Other Names: Global Quality of Recovery-40 score; Standard Pain Follow up and Monitorization
  Arms: Group TLIP
Procedure: ESPB — Patients will receive ESPB with an injection of 40 ml of bupivacaine 0.25% (2 injections of 20 ml on each side) between erector spinae muscle and transverse process of a vertebra.
  Other Names: Global Quality of Recovery-40 score; Standard Pain Followup and Monitorization
  Arms: Group ESP

SUMMARY:
Major spinal surgery causes greater pain in the postoperative 24 hours. Patients with severe pain may have prolonged hospital stays and delay in mobilization. In addition, chronic pain may be seen in these patients due to ineffectively managed acute postoperative pain. Therefore, optimizing acute postoperative analgesia is a priority in patients undergoing major spinal surgery.

Recently, ultrasound-guided interfascial plane blocks such as thoracolumbar interfascial plane block (TLIPB)and the erector spinae plane block (ESPB) have been described in spinal surgery. Both blocks clinically seem to be safe and easily performed. The aims of this study are to compare the quality of recovery scores, overall morbidity and postoperative analgesia after major spinal surgery in patients receiving either TLIPB or ESPB.

DETAILED DESCRIPTION:
Thoracolumbar interfascial plane block (TLIPB)and erector spinae plane block (ESPB) and have been shown to provide effective analgesia after spinal surgery. ESPB targets ventral and dorsal rami of the spinal nerve and also spreads over the paravertebral and epidural space. However, TLIPB targets only dorsal rami of the spinal nerve and spare ventral rami which may provide early ambulation. In addition, depositing local anesthetic in the fascial planes may prevent intraoperative washout. It may translate to an increase in the quality of analgesia. On the other hand, pain is an incomplete measure of postoperative recovery. No study to date has compared these two blocks in terms of the quality of recovery after major spinal surgery. This study will test the hypothesis that patients receiving TLIPB have higher QoR-40 scores in comparison with patients receiving ESPB.

ELIGIBILITY:
Inclusion Criteria:

-≥ 18 years old,

* Undergoing posterior lumbar spinal one to three levels fusion surgery
* Having signed a written informed consent form,
* ASAI-III

Exclusion Criteria:

* Contraindication for regional anesthesia (allergy to local anesthetics, neuropathic disease, infection at the puncture site, coagulation disorder, refusal of the technique,…)
* Contraindication to nonsteroidal anti-inflammatory drugs,
* Patient who has already had a spinal surgery,
* Patient with chronic pain syndrome (use > 3 months of morphine, opioid analgesics of class 3, pregabalin or gabapentin) or fibromyalgia,
* A mental or linguistic inability to understand the study,
* Pregnant or or breastfeeding women,
* Patient who can not communicate in Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (QoR-40) Score | Postoperative 24th hour
  QoR-40, a 40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain. I rate each item on a scale of 1-5, providing a minimum score of 40 and maximum of 200.QoR-40, a 40-item questionnaire that provides a global score and sub-scores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Each item is rated on a scale of 1-5, providing a minimum score of 40 and maximum of 200.Global QoR-40 scores range from 40 to 200 representing, respectively, very poor to outstanding quality of recovery. QoR-40 score will be recorded on the morning of operation and at the postoperative 24th hour.

SECONDARY OUTCOMES:
Area under the Numeric Rating Scale pain score versus time | Postoperative 24 hours
  11-point Numerical Rating Scale pain score is measured from '0' (means no pain) to '10' (means worst pain imaginable) both at rest and during sitting.
Numeric Rating Scale pain score | Postoperative 24 hours
  Pain scores using a Numeric Rating Scale (NRS) ranging from 0 to 10 (0= no pain; 10= worst imaginable pain). These scores will be recorded before surgery, in PACU and 6th, 12th and 24th at the postoperative period, both at rest and during sitting.
  and 24th hour pain imaginable).
Documentation of adverse events | Postoperative 24 hours
  Nausea and vomiting
Postoperative opioid consumption in the first 24 hours | Postoperative 24 hours
  Subjects will be extubated, taken to the postanesthesia care unit (PACU) and will be received by a nurse blinded to randomization. A standard PACU opioid algorithm will be used which involved:
  1. intravenous fentanyl 25 µg for Numeric Rating Scale (NRS) pain scores of either 4 or 5
  2. intravenous fentanyl 50 µg for NRS of 6 or greater. On discharge to the ward, subjects will be provided immediate-release oral oxycodone 5 mg every 4 hours as needed for NRS of 4-6; and 10 mg every 4 hours as needed for NRS of 7-10.
  All opioid doses will be converted to morphine equivalents.
Time for administration of first opioid analgesia | Postoperative 24 hours
  Time to administration of first opioid analgesia in the postanesthesia care unit
Postoperative complications | Postoperative thirty days
  Postoperative complications will be identified by visiting patients every day or alternate day during their in-hospital course, supplemented by patients' medical records review by assessors masked to group allocation, using our hospital's electronic patient record database. We will use the Claviene Dindo Classification system from which CCI is derived. We defined a postoperative complication as any deviation from the ideal postoperative course, not inherent in the procedure itself and does not constitute a failure to cure. CCI scores will be calculated using the online CCI calculator.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Basaran, MD, DESA, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)